CLINICAL TRIAL: NCT00824135
Title: Haploidentical Hematopoietic Stem Cell Transplantation Using A Novel Clofarabine Containing Conditioning Regimen For Patients With Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REFLEX; NCI-2011-03677 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Hematologic Malignancies
Keywords: Stem Cell Transplantation, Hematopoietic; Peripheral Blood Stem Cell Transplantation; Maximal Tolerated Dose; Clofarabine; Hematological Malignancies; Apheresis
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Clofarabine; Hematopoietic Stem Cell Transplantation; Muromonab-CD3; Thiotepa; Melphalan; Mycophenolic Acid; Rituximab; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Clofarabine; Procedure: Stem Cell Transplantation, Hematopoietic; Other: OKT3; Drug: Thiotepa; Drug: Melphalan; Drug: Mycophenolate mofetil; Drug: Rituximab; Other: G-CSF

INTERVENTIONS:
Drug: Clofarabine — One dose intravenously every 24 hrs for five days total.
  Dose level 1 Clofarabine 40 mg/m2/day intravenous Dose level 2 Clofarabine 45 mg/m2/day intravenous Dose Level 3 Clofarabine 50 mg/m2/day intravenous
Procedure: Stem Cell Transplantation, Hematopoietic — Haploidentical Hematopoietic Stem Cell Transplantation (two infusions, one on day 0 and the other on day +1)
Other: OKT3 — Start at 0.0125 mg/kg intravenous once a day, taper dose down incrementally and discontinue after 17 days total
  Muromonab-CD3
  Other Names: Orthoclone OKT3
Drug: Thiotepa — 5 mg/kg/day intravenous every 12 hours (2 doses total)
Drug: Melphalan — 60mg/m2 intravenous every 12 hours for 2 doses total.
Drug: Mycophenolate mofetil — Mycophenolate mofetil 600 mg/m2 intravenous two times a day
  (continue for approximately 2 months or as clinically indicated)
  Other Names: MMF; CellCept
Drug: Rituximab — 375 mg/m2 intravenous for 1 dose total
  Other Names: Rituxin
Other: G-CSF — G-CSF 5 mcg/kg/day subcutaneous or intravenous until ANC greater than 2.000/mm3 for 2 consecutive days and then as clinically indicated.

SUMMARY:
Patients with refractory hematologic malignancies including those who develop recurrent disease after allogeneic hematopoietic stem cell transplantation (HSCT) have a dismal prognosis. Historically, both regimen-related mortality and disease recurrence have been significant causes of treatment failure in this heavily pre-treated patient population. The investigators institution has utilized mismatched family member donors for these patients for several reasons: (1) Only 30% of patients have matched related donors available; (2) transplantation can be performed more rapidly since the time to unrelated donor trans-plantation averages 3 to 4 months; (3) the alloimmune reactivity of natural killer (NK) cells following haploidentical HSCT has been shown to reduce relapse rates in certain patient groups; and, (4) no other curative treatment options are available.

In the present trial, the investigators propose a novel conditioning regimen using clofarabine in an effort to enhance cytotoxicity while simultaneously reducing regimen related toxicity. In this phase I trial, the goal is to determine the maximum tolerated dose (MTD) of clofarabine when used in combination with melphalan and thiotepa pre-transplant.

DETAILED DESCRIPTION:
The primary objective of this trial is to determine the maximum tolerated dose of clofarabine in combination with thiotepa and melphalan as a conditioning regimen for a haploidentical stem cell transplant with an engineered graft depleted of CD3+ cells. Study participants will children and young adults with refractory hematologic malignancies.

Secondary objectives include the following:

* To describe the one-year overall survival (OS) and event-free survival (EFS) rates in these study participants.
* To determine the time to hematopoietic recovery and donor cell engraftment following this study treatment.
* To estimate the cumulative incidence of relapse in study participants.
* To estimate the incidence of overall grade II-IV and grade III-IV acute GVHD and the rate of chronic GVHD.
* To estimate the incidence and describe the causes of non-hematologic regimen-related toxicity and regimen-related mortality in the first 100 days post HSCT.
* To explore the biologic significance of soluble interleukin-2 (IL-2) receptor, tumor necrosis factor (TNF), and lymphocyte reconstitution (qualitative and quantitative, V beta spectratyping, TREC

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 21 years old; may be greater than 21 years old if a previously treated St. Jude patient and within 3 years of completion of most recent prior disease specific therapy.
* One of the following refractory hematologic malignancies (chemoresistant relapse or primary induction failure) or diagnoses:
* ALL
* AML (>25% blasts in the bone marrow)
* secondary AML/MDS
* CML in accelerated phase or blast crisis
* juvenile myelomonocytic leukemia (JMML)
* myelodysplastic syndrome (MDS)
* Hodgkin or non-Hodgkin lymphoma (NHL) with residual or recurrent disease following autologous HSCT, who are unable to undergo autologous HSCT due to chemo-resistant disease or inability to have an acceptable quantity of tumor-free stem cells collected (> 1 x 108 TNC/kg marrow or > 1 x 106 CD34+/kg PBS
* patients with a hematologic malignancy who have undergone prior allogeneic HSCT or who have a co-morbid condition that in the medical opinion of medical faculty (Division of Bone Marrow Transplantation and Cellular Therapy) makes standard myeloablation prohibitive
* Does not have any other active malignancy other than the one for which this transplant is indicated
* Cardiac shortening fraction greater than or equal to 25%
* For pediatric patients, creatinine clearance greater than or equal to 90 ml/min/1.73 m2 according to the Schwartz formula for estimated GFR (ml/min/1.73m2) = k*height (cm)/serum creatinine (mg/dL). k is a proportionality constant that varies with age and is a function of urinary creatinine clearance per unit of body size; 0.45 up to 12 months of age; 0.55 children and adolescent girls; and 0.70 for adolescent boys
* For adolescent or adult patients, serum creatinine 1.0 mg/dL; if serum creatinine 1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be 60 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation where predicted GFR (ml/min/1.73 m2) = 186 x (serum creatinine)-1.154 x (age in years)-0.023 x (0.742 if patient is female) x (1.212 if patient is black)
* Forced vital capacity (FVC) greater than or equal to 40% of predicted value or pulse oximetry greater than or equal to 92% on room air.
* Karnofsky or Lansky (age-dependent) performance score of greater than or equal to 50 (See APPENDIX A)
* Does not have active acute or active chronic GVHD defined as requiring medical therapy.
* Does not have active acute bronchiolitis obliterans (BO) or bronchiolitis obliterans organizing pneumonia (BOOP).
* Has a suitable HLA partially matched family member donor available for stem cell donation
* Bilirubin less than or equal to 1.5 times the upper limit of normal for age.
* Alanine aminotransferase (ALT) less than or equal to 1.5 times the upper limit of normal for age.
* Aspartate aminotransferase (AST) less than or equal to 1.5 times the upper limit of normal for age.
* Not pregnant (confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment).
* Not lactating

Inclusion criteria (stem cell donor):

* Partially HLA-matched family member.
* At least 18 years of age.
* HIV negative
* Not pregnant (confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment).
* Not lactating

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2009-01; Primary Completion 2012-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To determine the MTD and DLT of clofarabine in combination with thiotepa and melphalan as a conditioning regimen for a haploidentical HSCT with an engineered graft depleted of CD3+ cells obtained by negative selection with OKT3 on the CliniMACS system. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols